CLINICAL TRIAL: NCT03345667
Title: Assessment of Color Vision in Diabetic Patients Before and After the Use of Anti-vegf in the Treatment of Diabetic Macular Edema
Brief Title: Assessment of Color Vision in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: TRABALHO PEDRO ARVO 2018
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Retinopathy, Diabetic
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anti-Vegf: Use intravitreous anti-vegf
  Interventions: Drug: lucentis

INTERVENTIONS:
Drug: lucentis — Use of lucentis and other anti-vegf in patients with diabetic retinopathy

SUMMARY:
Assessment of color vision in diabetic patients before and after the use of anti-vegf in the treatment of diabetic macular edema

ELIGIBILITY:
Inclusion Criteria:

* Having diabetic retinopathy with macular edema

Exclusion Criteria:

* Not having diabetic retinopathy with macular edema

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Assessment of color vision in diabetic patients before and after the use of anti-vegf in the treatment of diabetic macular edema. Using the Ishirara's test to evaluate the possible visual loss.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Assessment of color vision in diabetic patients before and after the use of anti-vegf in the treatment of diabetic macular edema | 3 months
  Using the Ishihara's test to analise the possible loss of vision

SECONDARY OUTCOMES:
Frame between the injections | 1 months
  Ant-Vegf

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No